CLINICAL TRIAL: NCT05972655
Title: Modified Short-Course Radiation Combined With CAPOX and Tislelizumab for MSS Locally Advanced of Middle and Low Rectal Cancer (mRCAT): An Open-label, Single-arm, Prospective Multicenter Clinical Trial
Brief Title: Nodes-sparing Short-course Radiation Combined With CAPOX and Tislelizumab for MSS Middle and Low Rectal Cancer
Acronym: mRCAT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRRS-mRCAT
Record Dates: First submitted 2023-07-20; First posted 2023-08-02 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Low Rectal Cancer
MeSH Terms: interventions — spartalizumab; Capecitabine; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): Participants will receive 5*5Gy modified short-course radiation (radiation targeting the tumor bed without irradiating surrounding tumor-draining lymph nodes) concurrently with CAPOX and tislelizumab regimens: Oxaliplatin, 130mg/m2, intravenous infusion,d1 of each cycle; Capecitabine, 1000mg/m2, PO, BID, d1-14 and tislelizumab, 200mg intravenous infusion d1 of each cycle. CAPOX and tislelizumab repeat every 3 weeks for 4 cycles, followed by total mesorectal excision surgery.
  Interventions: Radiation: Modified short-course radiotherapy; Drug: PD-1 antibody; Drug: Capecitabine; Drug: Oxaliplatin

INTERVENTIONS:
Radiation: Modified short-course radiotherapy — radiation targeting the tumor bed without irradiating surrounding tumor-draining lymph nodes: 25Gy/5Fx
Drug: PD-1 antibody — PD-1 antibody (Tislelizumab): 200mg d1 q3w
Drug: Capecitabine — Capecitabine: 1000mg/m2 d1-14 q3w
Drug: Oxaliplatin — Oxaliplatin: 130mg/m2 d1 q3w

SUMMARY:
This is an open-label, prospective, multicenter phase II clinical trial to evaluate modified short-course radiation (Radiation targeting the tumor bed without irradiating surrounding tumor-draining lymph nodes) combined with CAPOX and PD-1 Inhibitor (Tislelizumab) for patients with MSS middle and low rectal cancer. A total of 32 patients will be enrolled in this trial. The primary endpoint is the rate of pathological complete response (pCR). The organ preservation rate, tumor regression grade, long-term prognosis, and adverse effects will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a strong willingness to preserve the anus and are willing to receive neoadjuvant therapy.
2. Male or Female aged 18-75.
3. Patients diagnosed with low rectal cancer within 10 cm from the lower edge of the tumor to the anal verge by pelvic MRI and anorectoscopy, the clinical stage is cT2N+M0/cT3-4aN0/+M0, the lymph nodes are limited to the mesorectum, the circumferential resection margin is negative.
4. Histologically confirmed rectal adenocarcinoma; Genetic testing suggests MSI-L or MSS, or tumor biopsy immunohistochemistry reveals pMMR, that is, MSH1, MSH2, MSH6, and PMS2 are all positive.
5. Eastern Cooperative Oncology Group (ECOG) 0-1.
6. No previous treatment(including anti-tumor therapy、immunotherapy or pelvic radiation).
7. Adequate hematologic, hepatic, renal, thyroid and cardiac function: white blood cells ≥3500/mm3, neutrophils ≥1800/mm3, platelets ≥100,000/mm3, hemoglobin ≥100 g/L; activated partial thromboplastin time, prothrombin time and international normalized ratio ≤1.5 × ULN; aspartate aminotransferase and alanine aminotransferase ≤3.0 × upper limit of normal (ULN), bilirubin ≤1.25 × ULN, serum albumin ≥28 g/L. creatinine clearance ≥50 mL/mi, creatinine ≤1.5 × ULN;
8. Informed consent form signed.

Exclusion Criteria:

1. Patients with a previous history of malignant tumors besides rectal cancer.
2. Patients with distant metastases before enrollment.
3. Patients with positive internal or external iliac lymph nodes are assessed by MRI or CT.
4. Patients with obstruction, perforation, or bleeding that require emergency surgery.
5. Patients with severe concomitant diseases and estimated survival time ≤ 5 years.
6. Allergic to any component of the therapy.
7. Patients with poorly differentiated adenocarcinoma, signet ring cell carcinoma, or mucinous adenocarcinoma.
8. Patients who received immunosuppressive or systemic hormone therapy for immunosuppressive purposes within 1 month prior to the initiation of therapy.
9. Patients who have received any other experimental drug (including immunotherapy) or participated in another interventional clinical trial within 30 days before screening.
10. Factors leading to study termination, such as alcoholism, drug abuse, other serious illnesses (including psychiatric disorders) requiring combination therapy, and patients with severe laboratory abnormalities.
11. Patients with congenital or acquired immune deficiency (such as HIV infection).
12. Vulnerable groups, including mentally ill, cognitively impaired, critically ill patients, minors, pregnant or lactating women, illiterate, etc.
13. Other conditions that investigators consider not suitable for this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | within 10 days after surgery
  The status of pCR will be evaluated after the TME surgery.

SECONDARY OUTCOMES:
Tumor regression grade | within 10 days after surgery
  TRG is evaluated according to the AJCC system. TRG0-1 is defined as good response, TRG2 as moderate response, and TRG3 as poor response.
Local recurrence rate(LRR) | 3 years after sugery
  Presence of adenocarcinoma within the rectal wall or within the mesorectum confirmed by pathology.
Disease free survival(DFS) | 3 years after surgery
  The three-year disease-free survival of patients.
Overall survival(OS) | 3 years after surgery
  The three-year overall survival of patients.
Adverse effects rate | From date of initiation of treatment until the date of death from any cause, assessed up to 5 years
  Rate of radiotherapy, chemotherapy and immunotherapy related adverse events
Rectal specific quality of life assessment via QLQ-CR29 | Baseline and months 3, 6, 12, 24, 36, 60 after the surgery
  Rectal specific quality of life according to European Organization for Research and Treatment of Cancer ( EORTC) Quality of life questionnaire QLQ-CR29. scale from 0 to 100, A higher scale represents better function and a higher quality of life.
Quality of life assessment via QLQ-C30 | Baseline and months 3, 6, 12, 24, 36, 60 after the surgery
  Quality of life according to EORTC Quality of life Questionnaire QLQ-C30 version 3.0. Score range from 0 to 100 points. A higher score represents better function and a higher quality of life.
Validation of the Wexner score | Months 3, 6, 12, 24, 36, 60 after the surgery
  The change of severity of fecal incontinence assessment according to Wexner score. a score from 0-20, where 0 is perfect continence and 20 is complete incontinence.

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Run Run Shao hospital, Hanzhou, Zhejiang, China

REFERENCES:
- [Derived] Cai C, Zhang X, Sun X, Wang H, Chen E, Chen L, Gu B, Wang J, Huang X, Lao W, Wang X, Chen M, Ding S, Du J, Song Z. Node-sparing modified short-course Radiotherapy Combined with CAPOX and Tislelizumab for locally Advanced MSS of Middle and low rectal Cancer (mRCAT): an open-label, single-arm, prospective, multicentre clinical trial. BMC Cancer. 2024 Oct 9;24(1):1247. doi: 10.1186/s12885-024-12994-0. PMID 39385104